CLINICAL TRIAL: NCT00200499
Title: A Multi-Center, Parallel Group Extension Study to Determine the Safety and Efficacy of Long-Term Nebivolol Exposure in Patients With Mild to Moderate Hypertension
Brief Title: A Study of the Safety and Efficacy of Long-Term Nebivolol Use in Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Bertek Pharmaceuticals (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NEB306
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-12-16 (Estimated); Status verified 2005-09

CONDITIONS: Hypertension
Keywords: Nebivolol; Hypertension; Beta-Blocker
MeSH Terms: conditions — Hypertension | interventions — Nebivolol

INTERVENTIONS:
Drug: Nebivolol

SUMMARY:
The study was conducted to determine the long-term safety and efficacy of nebivolol in patients with mild to moderate hypertension. This was an extension of the Phase III dose ranging studies NEB 202, 302 and 305. Nebivolol was studied as monotherapy and in conjunction with add-on antihypertensive therapy.

DETAILED DESCRIPTION:
This was an international, multicenter parallel group, 9-month extension study with a 4-week follow-up phase to evaluate the long-term safety and efficacy of nebivolol administered orally once daily in patients with mild to moderate hypertension (defined as an average sitting diastolic blood pressure greater then or equal to 95 mmHg and less then or equal to 109 mmHg when untreated, based on entry into NEB 202, NEB 302 or NEB 305). Patients were permitted protocol-defined concomitant use of diuretic or calcium antagonist. After successful completion of one of the 3-month efficacy "feeder" studies, patients were eligible to continue nebivolol treatment in this 9-month extension study. Patients who completed the extension phase and received only nebivolol monotherapy during the extension phase were eligible to enter the 1-month follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* To enter the long-term treatment phase, patients must have successfully completed NEB 202, NEB 302, or NEB 305. To enter the 4-week follow-up phase, patients must have completed NEB-306 (extension phase) and received only nebivolol monotherapy treatment during NEB 306.

Exclusion Criteria:

* Secondary hypertension
* myocardial infarction or stroke
* contraindications to beta-blocker therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 845
Dates: Start 2002-03; Study Completion 2003-09

PRIMARY OUTCOMES:
The change in average sitting diastolic blood pressure measured at trough drug plasma level at the end of the extension phase compared to baseline of NEB 202, NEB 302 or NEB 305.

SECONDARY OUTCOMES:
Change in the average
- sitting systolic blood pressure
- supine and standing systolic and diastolic blood pressure
- response rate of treatment groups
- AEs
- ECGs
- laboratory parameters
- heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Betty S. Riggs, MD, MBA, Study Director — Mylan Pharmaceuticals Inc
Locations (1):
- Mylan Pharmaceuticals Inc., Morgantown, West Virginia, United States